CLINICAL TRIAL: NCT02634164
Title: The Effects of Leucine and Isoleucine on Glucose Metabolism
Acronym: AA+GLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17757
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Hyperglycemia
Keywords: leucine; isoleucine
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- control (No Intervention): Control Treatment with Oral Glucose Tolerance Test:
  Blood glucose and insulin will be obtained following the protocol of Eicher et al (4). Participants will ingest a Placebo (inert, calorie free, stevia sweetener) with blood collections at 0,2,4,6,8,10,30 prior to a standard 75 g glucose solution, followed by blood collections at 0,2,4,6,8,10,30,60,90,120 minutes post glucose ingestion. A total of 16 blood collections will be taken.
- Leucine Supplement (Experimental): Control Treatment with Oral Glucose Tolerance Test:
  Interventions: Dietary Supplement: Leucine Supplement
- Isoleucine Supplement (Experimental): Isoleucine Combined with Oral Glucose Tolerance Test:
  Interventions: Dietary Supplement: Isoleucine Supplement
- Leucine and Isoleucine Supplement (Experimental): Leucine and Isoleucine Combined with Oral Glucose Tolerance Test:
  Interventions: Dietary Supplement: Leucine Supplement combined with Isoleucine Supplement

INTERVENTIONS:
Dietary Supplement: Leucine Supplement — For this visit participants will ingest a powdered form of Leucine in the amount of 0.3g/kg of lean body mass weight with water (150 mL) with additional water if needed to ensure dose is fully consumed. The amino acid solution will be ingested 30 min prior to 75 g glucose solution
  Arms: Leucine Supplement
Dietary Supplement: Isoleucine Supplement — For this visit participants will ingest a powdered form of Isoleucine in the amount of 0.3g/kg of lean body mass weight with water (150 mL) with additional water if needed to ensure dose is fully consumed. The amino acid solution will be ingested 30 min prior to 75 g glucose solution.
  Arms: Isoleucine Supplement
Dietary Supplement: Leucine Supplement combined with Isoleucine Supplement — For this visit participants will ingest a powdered form of Leucine and Isoleucine in the amount of 0.3g/kg of lean body mass weight (equal in total dosage to other treatments) with water (150 mL) with additional water if needed to ensure dose is fully consumed. The amino acid solution will be ingested 30 min prior to 75 g glucose solution.
  Arms: Leucine and Isoleucine Supplement

SUMMARY:
Diabetes is classified as an impairment of the body's ability to control blood glucose levels. Uncontrolled hyperglycemia can give rise to macrovascular (i.e., heart disease and stroke) and microvasculature damage such as retinopathy, nephropathy and neuropathy. These comorbidities may definitively reduce quality of life.

Hypotheses to be tested:

1. The ingestion of amino acids L-Isoleucine and L-Leucine at a therapeutic dose prior to a glucose load will concurrently and independently improve glucose tolerance.
2. The ingestion of L-Isoleucine and L-Leucine separately or together will have a minimal effect on incretin responses of Glucagon-like peptide-1 and Glucose-dependent insulinotropic peptide (GLP-1, GIP).

DETAILED DESCRIPTION:
Specific Aims and Hypothesis Diabetes is classified as an impairment of the body's ability to control blood glucose levels. Uncontrolled hyperglycemia can give rise to macrovascular (i.e., heart disease and stroke) and microvasculature damage such as retinopathy, nephropathy and neuropathy. These comorbidities may definitively reduce quality of life.

Hypotheses to be tested:

1. The ingestion of amino acids L-Isoleucine and L-Leucine at a therapeutic dose prior to a glucose load will concurrently and independently improve glucose tolerance.
2. The ingestion of L-Isoleucine and L-Leucine separately or together will have a minimal effect on incretin responses (GLP-1, GIP).

Specific Aims:

1. Specific Aim I will test the hypothesis that the ingestion of amino acids L-Isoleucine and L-Leucine at a therapeutic dose prior to a glucose load will concurrently and independently improve glucose tolerance.
2. Specific Aim II will test the hypothesis that the ingestion of L-Isoleucine and L-Leucine will have a minimal effect on incretin responses in conjunction with prior research.

ELIGIBILITY:
Inclusion Criteria:

1. age range of 20 to 40 years of age
2. (sedentary lifestyle) Participants whom exercise less than the American College of Sports Medicine recommendation of weekly physical activity levels or are completely sedentary may be admitted into the study
3. Apparently healthy
4. Currently not using supplemental branch chain amino acids (BCAA) or whey protein
5. Non-smoking

Exclusion Criteria:

1. Chronic or acute health problems
2. Smoker
3. Currently using supplemental BCAA or whey protein -

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood collections
Change in plasma insulin (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood collections
Change in plasma GIP (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood Collections
Change in plasma GLP-1 (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood collections

SECONDARY OUTCOMES:
Change in plasma glucagon (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood collections
Change in plasma c-peptide (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood Collections
Change in plasma L-Leucine (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood Collections
Change in plasma L-Isoleucine (0-150 minutes) | baseline (0), 2, 4, 6, 8, 10, 30, 32, 34, 36, 38, 40, 60, 90, 120, 150 minutes
  Blood Collections

CONTACTS AND LOCATIONS:
Overall Officials: Vic Ben-Ezra, PhD, Study Chair — Texas Woman's University Kinesiology Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshizawa F. New therapeutic strategy for amino acid medicine: notable functions of branched chain amino acids as biological regulators. J Pharmacol Sci. 2012;118(2):149-55. doi: 10.1254/jphs.11r05fm. Epub 2012 Jan 27. PMID 22293293
- [Result] Nuttall FQ, Schweim KJ, Gannon MC. Effect of orally administered phenylalanine with and without glucose on insulin, glucagon and glucose concentrations. Horm Metab Res. 2006 Aug;38(8):518-23. doi: 10.1055/s-2006-949523. PMID 16941278
- [Result] Gannon MC, Nuttall FQ. Amino acid ingestion and glucose metabolism--a review. IUBMB Life. 2010 Sep;62(9):660-8. doi: 10.1002/iub.375. PMID 20882645
- [Result] Kalogeropoulou D, Lafave L, Schweim K, Gannon MC, Nuttall FQ. Leucine, when ingested with glucose, synergistically stimulates insulin secretion and lowers blood glucose. Metabolism. 2008 Dec;57(12):1747-52. doi: 10.1016/j.metabol.2008.09.001. PMID 19013300
- [Result] Nilsson M, Holst JJ, Bjorck IM. Metabolic effects of amino acid mixtures and whey protein in healthy subjects: studies using glucose-equivalent drinks. Am J Clin Nutr. 2007 Apr;85(4):996-1004. doi: 10.1093/ajcn/85.4.996. PMID 17413098
- [Result] Petersen BL, Ward LS, Bastian ED, Jenkins AL, Campbell J, Vuksan V. A whey protein supplement decreases post-prandial glycemia. Nutr J. 2009 Oct 16;8:47. doi: 10.1186/1475-2891-8-47. PMID 19835582
- [Result] Doi M, Yamaoka I, Fukunaga T, Nakayama M. Isoleucine, a potent plasma glucose-lowering amino acid, stimulates glucose uptake in C2C12 myotubes. Biochem Biophys Res Commun. 2003 Dec 26;312(4):1111-7. doi: 10.1016/j.bbrc.2003.11.039. PMID 14651987
- [Result] Nishitani S, Takehana K, Fujitani S, Sonaka I. Branched-chain amino acids improve glucose metabolism in rats with liver cirrhosis. Am J Physiol Gastrointest Liver Physiol. 2005 Jun;288(6):G1292-300. doi: 10.1152/ajpgi.00510.2003. Epub 2004 Dec 9. PMID 15591158